CLINICAL TRIAL: NCT00517868
Title: URG101 Pharmacodynamic and Safety Study: A Randomized, Double-blind, Placebo-controlled, Multi-center Cross-over Study to Investigate the Pharmacodynamic Profile of URG101 in Subjects With Pelvic Pain of Bladder Origin.
Brief Title: Study of URG101 in Painful Bladder Syndrome and Interstitial Cystitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to Food and Drug Administration (FDA) recalled the heparin used in the trial because of possible contamination.
Sponsor: Urigen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: URG101-104
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Results first posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Painful Bladder Syndrome; Interstitial Cystitis; Bladder Pain Syndrome
Keywords: bladder; pain; urgency; frequency
MeSH Terms: conditions — Cystitis, Interstitial; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crossover (Other): Placebo Treatment on Visit 1 followed by URG101 Treatment on Visit 2
  Interventions: Drug: URG101; Drug: Placebo
- Crossover 2 (Other): URG101 Treatment on Visit 1 followed by Placebo Treatment on Visit 2
  Interventions: Drug: URG101; Drug: Placebo

INTERVENTIONS:
Drug: URG101 — Bladder instillation of URG101 or Placebo in random order on treatment 1 and treatment 2 followed by an open-label URG101 on treatment 3 within the same week.
Drug: Placebo — Liquid formulation without active URG101 drug components

SUMMARY:
A double-blind, placebo-controlled study to evaluate changes in pain, urgency and urinary frequency following administration of URG101 compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* male and female subjects >= 18 years of age
* moderate to severe symptoms of PBS/IC
* minimum pain/urgency/frequency scores
* female subjects on hormone therapy must be on stable dose for >= 3 months

Exclusion Criteria:

* positive pregnancy test or pregnant or lactating
* narcotics or medical marijuana within 3 months
* use of any investigational drug or device within 30 days
* bacterial cystitis within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-08-28 (Actual); Primary Completion 2008-02-28 (Actual); Study Completion 2008-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Proctor, M.D., Principal Investigator — Georgia Urology
Locations (6):
- United States (6):
  - Citrus Valley Medical Research, Glendora, California
  - SD Uro-Research, San Diego, California
  - University of California, San Diego, San Diego, California
  - Scripps Clinic Medical Group, San Diego, California
  - Georgia Urology, Cartersville, Georgia
  - Urology San Antonio Research, P.A., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parsons CL, Zupkas P, Proctor J, Koziol J, Franklin A, Giesing D, Davis E, Lakin CM, Kahn BS, Garner WJ. Alkalinized lidocaine and heparin provide immediate relief of pain and urgency in patients with interstitial cystitis. J Sex Med. 2012 Jan;9(1):207-12. doi: 10.1111/j.1743-6109.2011.02542.x. Epub 2011 Nov 14. PMID 22082303

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 28 participants received at least one dose in both Crossover Group 1 and Crossover Group 2. A third arm, All Dosed Subjects, has been listed to the Participant Flow section to allow for overall study Baseline Characteristics to be entered.
Groups:
- Crossover Group 1: Placebo Treatment on Visit 1 followed by URG101 Treatment on Visit 2
  URG101: Bladder instillation of URG101 or Placebo in random order on treatment 1 and treatment 2 followed by an open-label URG101 on treatment 3 within the same week.
  Placebo: Liquid formulation without active URG101 drug components
- Crossover Group 2: URG101 Treatment on Visit 1 followed by Placebo Treatment on Visit 2
  URG101: Bladder instillation of URG101 or Placebo in random order on treatment 1 and treatment 2 followed by an open-label URG101 on treatment 3 within the same week.
  Placebo: Liquid formulation without active URG101 drug components
Period: Overall Study
Arm/Group | Crossover Group 1 | Crossover Group 2
Started | 18 | 10
Completed | 16 | 10
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Population: Subjects randomized per crossover arm as of the time of study termination.
Groups:
- All Participants Dosed: Includes all participants who received at least one dose of URG101 or Placebo
  (Placebo: Liquid formulation without active URG101 drug)
Arm/Group | All Participants Dosed
Number analyzed (Participants) | 28
Age, Customized [Count of Participants; unit: Participants]
  ≥18 years of age | 28
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 1
  Female | 17
  Unknown | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 28

OUTCOME MEASURES:

1. Primary Outcome: Change in Daytime Bladder Pain Intensity
Description: A calculation of average bladder pain intensity differences from baseline to 12 hours post-dose , as determined using an 11-point numerical rating scale (NRS) for bladder pain from time of dosing through 12 hours post dose. The 11-point NRS for bladder pain is a scale from 0 to 10, with 0 indicating no bladder pain and 10 indicating the worst imaginable bladder pain.
Time Frame: Through 12 hours
Population: Subjects included in this analysis must have received at least the first two dose administrations and must have been determined to be evaluable per the Statistical Analysis Plan.
Measure: Mean (95% Confidence Interval); unit: Percentage of pain scale change
Groups:
- Placebo: Inclusive of all subjects who received at least one placebo dose as either the first or second dose administration.
- URG101: Inclusive of all subjects who received at least one URG101 (study drug) dose as either the first or second dose administration.
Arm/Group | Placebo | URG101
Number analyzed (Participants) | 18 | 18
Percentage of pain scale change | 20.73 [5.04 to 36.41] | 41.86 [27.64 to 56.08]
Statistical Analysis 1: Comparison: Placebo vs URG101; Test type: Non-Inferiority — A paired student t comparison was used to assess treatment differences as measured by 11 point numerical rating scale; p = 0.0363, t-test, 1 sided; Mean Difference (Final Values) = -21.14, 95% CI 2-sided [-44.43 to 2.16]

2. Secondary Outcome: Change in Question 3 of the Patient Overall Rating of Improvement of Symptoms (PORIS) Questionnaire
Description: Percentage of subjects achieving ≥ 50% improvement in Question 3 of the PORIS questionnaire at 12 hours post-dose. The PORIS questionnaire is an assessment of the subject's condition after treatment compared to before treatment. In particular, Question 3 of the PORIS questionnaire asks subjects to select the category that best describes the overall change in their condition compared to before receiving study medication; the choices are: worse, no better (0% improvement), slightly improved (25% improvement), moderately improved (50% improvement), greatly improved (75% improvement), or symptoms gone (100% improvement).
Time Frame: Through 12 hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | URG101
Number analyzed (Participants) | 18 | 18
Participants | 2 | 9

3. Secondary Outcome: Change in Total Symptom Score
Description: A calculation of the average percentage change of Total Symptom Score (including Pelvic/Bladder Pain and Urinary Urgency scales) differences from baseline to 12 hours post-dose, as determined using 11-point numerical rating scales (NRS) for Pelvic/Bladder Pain and Urinary Urgency from time of dosing through 12 hours post dose. The 11-point NRS for Pelvic/Bladder Pain is a scale from 0 to 10, with 0 indicating 'none' and 10 indicating the 'worst ever'. The 11-point NRS for Urinary Urgency (pressure to urinate) is a scale from 0 to 10, with 0 indicating 'none' and 10 indicating the 'worst ever'.
Time Frame: Through 12 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo | URG101
Number analyzed (Participants) | 18 | 18
Percentage of change | 17.04 (29.87) | 38.31 (27.73)

4. Secondary Outcome: Change in Daytime Urinary Urgency Score
Description: A calculation of average percentage change of Urinary Urgency differences from baseline to 12 hours post-dose, as determined using 11-point numerical rating scales (NRS) for Urinary Urgency from time of dosing through 12 hours post dose. The 11-point NRS for Urinary Urgency (pressure to urinate) is a scale from 0 to 10, with 0 indicating 'none' and 10 indicating the 'worst ever'.
Time Frame: Through 12 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Placebo | URG101
Number analyzed (Participants) | 18 | 18
Percentage of change | 13.30 (30.53) | 34.50 (30.21)

5. Post Hoc Outcome: Determination of Serum Lidocaine Levels Post Study Drug Administration
Description: Single-timepoint serum lidocaine measure at one hour following intravesical study drug administration
Time Frame: 1 hour post-dose
Population: Subjects who received at least one dose of URG101 and met protocol and statistical analysis plan criteria to be deemed evaluable.
Measure: Mean (Full Range); unit: µg/mL
Groups:
- Evaluable URG101 Subjects: Subjects who received at least one dose of URG101 and met protocol and statistical analysis plan criteria to be deemed evaluable.
Arm/Group | Evaluable URG101 Subjects
Number analyzed (Participants) | 18
µg/mL | 0.51 [0.24 to 2.0]

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) collection timeframe: for the duration of study conduct (up to 3 study visits or 5 days total) through 24 hours post-last dose of placebo or study drug Serious Adverse Event (SAE) and All-Cause Mortality (ACM) collection timeframe: for the duration of study conduct (up to 3 study visits or 5 days total) through 30 days post-last dose of placebo or study drug
Groups:
- Placebo: Inclusive of all AEs following placebo dose exposures.
- URG101: Inclusive of all AEs following URG101 (study drug) dose exposures.
- Total: Inclusive of all AEs following all placebo and URG101 dose exposures.
Arm/Group | Placebo | URG101 | Total
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28 | 1/28 | 1/28
Other Adverse Events (participants affected / at risk) | 8/28 | 21/28 | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=28) | URG101 (N=28) | Total (N=28)
Vaginal Bleeding (Reproductive system and breast disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=28) | URG101 (N=28) | Total (N=28)
Headache (Nervous system disorders) | 3 | 5 | 8
Dizziness (Nervous system disorders) | 1 | 2 | 3
Bladder Discomfort/Pain/Burning (Renal and urinary disorders) | 1 | 6 | 7
Urethral Pain/Burn/Discomfort (Renal and urinary disorders) | 1 | 1 | 2
Urinary Urgency (Renal and urinary disorders) | 1 | 1 | 2
Hematuria (Renal and urinary disorders) | 1 | 1 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 2 | 2
Vaginal Pain (Reproductive system and breast disorders) | 0 | 4 | 4

LIMITATIONS AND CAVEATS:
The study was intended to include 40 subjects, but it had to be terminated early because the Food and Drug Administration (FDA) unexpectedly recalled the heparin used in the trial due to a possible contamination.

Of the 28 subjects enrolled, limited demographic information is available, and the available data are reported for all subjects as a single group.

Of the 28 subjects enrolled, there were 18 evaluable full-crossover subjects for the statistical analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No